CLINICAL TRIAL: NCT06267521
Title: Hybrid Interventions to Optimize Neural Plasticity and Enhance Well-being: Mental Exercise, and Transcranial Electrical Stimulation With Temporal Interference: The STRENGTHEN Study - Phase 1 and 2
Brief Title: The STRENGTHEN Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2023-1473; Protocol Version 2/28/2025 (Other: UW Madison); L&S/PSYCHOLOGY/PSYCHOLOGY (Other: UW Madison); A487400 (Other: UW Madison); AWD00000302 (Other Grant/Funding Number: US Department of Defense DARPA)
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cognitive Flexibility; Emotional Regulation
MeSH Terms: conditions — Emotional Regulation | interventions — Transcranial Direct Current Stimulation; Neuroimaging

STUDY DESIGN:
Intervention Model Description: N= 48 into Phase 1, N=48 into Phase 2
Who Masked: Participant
Masking Description: Participants will not know whether they are in a group receiving active stimulation (groups 2, 3, and 4) or sham stimulation (group 1). However, participants will know whether they are performing meditation (groups 1, 3, and 4) or listening to only the didactic meditation material (group 2), and participants will be aware of how many nights they are undergoing stimulation (1 night per week for group 3, 2 nights per week for groups 1, 2, and 4). Thus, participants will be only partially blind to condition. Investigators will not be blind to condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Group 1: Mediation Only (Phase 1 and Phase 2) (Experimental): * Baseline measures including imaging
  * Meditation plus Sham Stimulation 2 nights per week for 4 weeks
  * Post Intervention (week 5) measures including imaging
  * Follow up measures (week 20)
  Interventions: Other: Healthy Minds Program; Device: Sham Stimulation in Lab; Device: MRI Scanner
- Group 2: Stimulation Only (Phase 1 and Phase 2) (Experimental): * Baseline measures including imaging
  * Sham Meditation plus Stimulation in Lab 2 nights per week for 4 weeks
  * Post Intervention (week 5) measures including imaging
  * Follow up measures (week 20)
  Interventions: Other: Sham Meditation Didactic Material; Device: Stimulation in Lab; Device: MRI Scanner
- Group 3: Combined, Low Frequency (Phase 1) (Experimental): * Baseline measures including imaging
  * Meditation plus Stimulation in Lab 1 night per week for 4 weeks
  * Post Intervention (week 5) measures including imaging
  * Follow up measures (week 20)
  Interventions: Other: Healthy Minds Program; Device: Stimulation in Lab; Device: MRI Scanner
- Group 4: Combined, High Frequency (Phase 1 and Phase 2) (Experimental): * Baseline measures including imaging
  * Meditation plus Stimulation in Lab 2 nights per week for 4 weeks
  * Post Intervention (week 5) measures including imaging
  * Follow up measures (week 20)
  Interventions: Other: Healthy Minds Program; Device: Stimulation in Lab; Device: MRI Scanner

INTERVENTIONS:
Other: Healthy Minds Program — Participants will follow daily instructions from the Healthy Minds Program at home for four weeks, including guided meditation exercises.
  Other Names: Health Minds App
  Arms: Group 1: Mediation Only (Phase 1 and Phase 2); Group 3: Combined, Low Frequency (Phase 1); Group 4: Combined, High Frequency (Phase 1 and Phase 2)
Other: Sham Meditation Didactic Material — Participants will listen to lessons from the Healthy Minds Program at home for four weeks, which will not include any actual meditation exercises.
  Arms: Group 2: Stimulation Only (Phase 1 and Phase 2)
Device: Sham Stimulation in Lab — On two nights each week during the four weeks of the intervention, participants will sleep in the lab and undergo sham TES-TI stimulation for approximately 10 hours per night
  Arms: Group 1: Mediation Only (Phase 1 and Phase 2)
Device: Stimulation in Lab — Participants will sleep in the lab and undergo active TES-TI stimulation for approximately 10 hours per night.
  Other Names: TES-TI; Transcranial Electrical Stimulation with Temporal Interference
  Arms: Group 2: Stimulation Only (Phase 1 and Phase 2); Group 3: Combined, Low Frequency (Phase 1); Group 4: Combined, High Frequency (Phase 1 and Phase 2)
Device: MRI Scanner — Imaging protocol will include: structural T1-weighted and T2-weighted images, resting-state functional MRI, task-based functional MRI, and multi-shell diffusion weighted MRI, total scan time will be approximately 2 hours
  Other Names: 3 Tesla MAGNUS; Microstructure Anatomy Gradient for Neuroimaging with Ultrafast Scanning

SUMMARY:
This study uses two different types of interventions including electrical brain stimulation delivered during sleep, and brief, daily meditation training. The investigators are trying to figure out whether these techniques, either alone or in combination with each other, can positively impact the brain networks that support our ability to think flexibly and to regulate our emotions. 48 participants will be enrolled into each of 2 phases and can expect to be on study for up to 9 months.

DETAILED DESCRIPTION:
The investigators will evaluate the independent and synergistic effect of Cognitive Flexibility (CF)/Emotional Regulation (ER) - targeted meditation and CF/ER-targeted Transcranial Electrical Stimulation with Temporal Interference (TES-TI) during sleep in low-risk participants (n = 48).

After informed consent, all participants will undergo a set of baseline assessments, including self-report measures, behavioral tasks, functional and structural MRI, and a baseline in-laboratory sleep study.

Following these assessments, participants undergo four weeks of the study intervention. The participants will be assigned into one of four groups. Each group consists of 12 participants.

After completing the 4-week intervention, participants will repeat the behavioral, self-report, and imaging assessments given at baseline. Participants will also complete a 7-day ecological momentary assessment (EMA) at baseline, the week after intervention, and at 4-months following intervention. At the 4-month follow-up, participants may complete another round of self-report and behavioral measures.

The Primary Objectives are to:

* Evaluate the effects of the following on CF and ER networks:

  1. meditation practice alone
  2. meditation practice and high-dose TES-TI
  3. meditation practice and low-dose TES-TI
  4. TES-TI alone

The Secondary Objectives are to:

* Evaluate the differential synergies between Non-Rapid Eye Movement (NREM) and Rapid Eye Movement (REM) sleep TES-TI intervention and the restoration of CF verses ER circuits

For Phase 2, an additional 48 participants will be recruited and will eliminate TES-TI once per week. All participants will come to the sleep laboratory for 2 nights over the 4 week intervention period.

Planned interim analysis of slow wave activity data from N=20 participants is adequately powered to evaluate whether TES-TI produces the anticipated modulation of deep sleep.

ELIGIBILITY:
Inclusion Criteria (Phase 1 and 2):

* Medically healthy
* English-speaking (able to provide consent and complete questionnaires)
* Citizen or legal resident

Exclusion Criteria (Phase 1):

* Any current or recent history (6 months) of any mental health diagnosis (Examples include major depression, hypomania, psychosis, schizophrenia, and bipolar disorder)
* Any current or recent (past 6 months) history of treatment for mental illness (including anti-depressant/anti anxiety medications, therapy)
* Scoring above Moderate range for Anxiety or Depression - Patient Health Questionnaire-9 (PHQ-9) greater than or equal to 15 or General Anxiety Disorder (GAD7) greater than or equal to 15
* At risk for suicide (PHQ item 9 greater than 0)
* Any current or past history of neurological disorders or acquired neurological disease (e.g. stroke, traumatic brain injury), including intracranial lesions and obstructive sleep apnea
* History of head trauma resulting in prolonged loss of consciousness; or a history of greater than 3 grade I concussions
* Current history of poorly controlled headaches including intractable or poorly controlled migraines
* Any systemic illness or unstable medical condition that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) electroencephalogram, or family history of treatment resistant epilepsy with the exception of a single seizure of benign etiology (e.g. febrile seizures) in the judgment of a board-certified neurologist
* Possible pregnancy or plan to become pregnant in the next 6 months.
* Any metal in the brain, skull or elsewhere
* Any hair braid, dreadlocks, hair pieces, or extensions which cannot be taken out before the MRI scans and/or sleep stimulation sessions
* Any head coverings or headdress that participant feels uncomfortable removing for the purposes of the MRI scans and/or sleep stimulation sessions
* Any medical devices or implants (i.e. cardiac pacemaker, medication infusion pump, cochlear implant, vagal nerve stimulator) unless otherwise approved by the responsible physician
* Dental implants containing metal (titanium or titanium alloys) surgically implanted post and core
* Substance use disorder within the past six months
* Any medication that may alter seizure threshold i.e., Attention-deficit/hyperactivity disorder (ADHD) stimulants (Adderall, amphetamine); Tricyclic/atypical antidepressants (amitriptyline, doxepine, imipramine, maprotiline, nortriptyline, bupropion); Antipsychotics (chlorpromazine, clozapine), Bronchodilators (theophylline, aminophylline); Antibiotics (fluoroquinolones, imipenem, penicillin, cephalosporins, metronidazole, isoniazid); Antivirals (valacyclovir, ritonavir); Over the Counter (OTC) (diphenhydramine, Benadryl)
* Claustrophobia (a fear of small or closed places)
* Back problems that would prevent lying flat for up to two hours
* Regular night-shift work (second or third shift)
* Do not have access to a smartphone or the internet
* Regular meditation practice and/or prior use of the Healthy Minds Program app
* Cannot visit the lab in-person for 7 consecutive weeks in the next year
* Permanent retainers

Additional Exclusion Criteria (Phase 2):

* Any current or recent history (6 months) of bipolar disorder, psychosis, schizophrenia. A history of stable depression or anxiety is not exclusionary.
* Mental health treatment (e.g, psychotherapy) is no longer exclusionary, although all the medication exclusions outlined above still apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ-9) Score | baseline, visit 3 (week 1), visit 4 (week 1), visit 5 (week 2), visit 6 (week 2), visit 7 (week 3), visit 8 (week 3), visit 9 (week 4), visit 10 (week 4), post-intervention (week 5), follow-up (week 20)
  The PHQ-9 is a 9-item inventory asking participants to rate from 0 (not at all) to 3 (nearly everyday) the frequency and intensity of depressive symptoms experienced by the respondent over the preceding two-week period. Scores range from 0 to 27 where higher scores indicate poorer patient health. Participants with scores greater than 15 will be excluded from study.
Change in General Anxiety Disorder (GAD-7) Score | baseline, visit 3 (week 1), visit 4 (week 1), visit 5 (week 2), visit 6 (week 2), visit 7 (week 3), visit 8 (week 3), visit 9 (week 4), visit 10 (week 4), post-intervention (week 5), follow-up (week 20)
  This 7-item inventory measures the severity of generalized anxiety disorder symptoms in individuals by asking participants to rate from 0 (not all at) to 3 (nearly everyday) the frequency and intensity of various anxiety-related symptoms experienced by the participant in the past two weeks. Scores range from 0-21 where higher scores indicate more anxiety. This study will exclude any participants who have a total score of 15 or above.
Change in Single-item Suicide Question | baseline, visit 3 (week 1), visit 4 (week 1), visit 5 (week 2), visit 6 (week 2), visit 7 (week 3), visit 8 (week 3), visit 9 (week 4), visit 10 (week 4), post-intervention (week 5), follow-up (week 20)
  This single-item suicide question assesses participant's suicidal ideation to respond yes or no to "Since the last time we saw you, did you seriously consider attempting suicide?".
Change in Healthy Minds Index (HM Index) | baseline, post-intervention (week 5), follow-up (week 20)
  The HM Index is a 17-question, 5-point scale well-being assessment that measures the four pillars of Wellbeing - Awareness, Connection, Insight, and Purpose. Means scores are from 1 to 5 with higher scores indicative of increased wellbeing.
Change in the Perceived Stress Scale (PSS) Score | baseline, post-intervention (week 5), follow-up (week 20)
  This is a 10-item inventory asking participants to rate from 0 (never) to 4 (very often) the frequency with which they have felt various kinds of stress in the last month. Scores range from 0 to 40 with higher score indicative of higher stress.
Change in Emotional Styles Questionnaire (ESQ) Score | baseline, post-intervention (week 5), follow-up (week 20)
  This is a 24-item inventory asking participants to rate from 1 (strongly disagree) to 7 (strongly agree). Scores range from 24 - 168, higher scores are indicative of less Healthy Emotionality
Change in Cognitive Flexibility Inventory (CFI) Score: Alternatives Subscale | baseline, post-intervention (week 5), follow-up (week 20)
  The CFI is a 20-item self-report measure to monitor how often individuals engage in cognitive behavioral thought challenging interventions. Participants rate each item from 1 (strongly disagree) to 7 (strongly agree). Scores range from 13 - 91, higher scores are indicative of increased ability to perceive multiple alternative explanations.
Change in Cognitive Flexibility Inventory (CFI) Score: Control Subscale | baseline, post-intervention (week 5), follow-up (week 20)
  The CFI is a 20-item self-report measure to monitor how often individuals engage in cognitive behavioral thought challenging interventions. Participants rate each item from 1 (strongly disagree) to 7 (strongly agree). Scores range from 7 - 49, higher scores are indicative of increased ability to perceive difficult situations as controllable.
Change in Difficulties in Emotion Regulation Scale-18 (DERS-18) Score | baseline, post-intervention (week 5), follow-up (week 20)
  The DERS-18 is a 18-item self-report measure which assesses various aspects of emotion regulation, including emotional awareness, acceptance of emotional responses, impulse control, and effective goal-directed behavior during emotional experiences using a 5-point scale from 1 (almost never) to 5 (almost always). Higher scores suggest greater problems with emotion regulation.
Change in PROMIS Sleep Disturbance Score | baseline, post-intervention (week 5), follow-up (week 20)
  This validated assessment tool asks participants to rate 8 items that measure sleep-related difficulties using a 5-point Likert scale. Scores range from 8 to 40 with higher scores indicative of more sleep disturbance.
Change in PTSD Checklist for DSM-5 (PCL-5) | baseline, post-intervention (week 5), follow-up (week 20)
  This 20-item self-report questionnaire is a widely used self-report questionnaire which assesses symptoms of post-traumatic stress disorder (PTSD). Participants rate from 0 (not at all) to 4 (extremely) the severity of their symptoms. Scores range from 0 to 80 with higher scores indicative of more severe PTSD symptoms.
Change in World Health Organization-5 (WHO-5) | baseline, post-intervention (week 5), follow-up (week 20)
  This 5-item scale is a global measure of Well-Being, where higher scores reflect greater overall wellbeing (range 0-25).
Change in Restorative Sleep Questionnaire (RSQ) Score | baseline, visit 3 (week 1), visit 4 (week 1), visit 5 (week 2), visit 6 (week 2), visit 7 (week 3), visit 8 (week 3), visit 9 (week 4), visit 10 (week 4)
  This validated assessment measuring subjective perceptions of the restorative or inadequate properties of sleep will be given the morning after every sleep lab visit. The questionnaire includes 9 items rated on a 5 point scale given at the time of awakening. Scores range from 0 to100, where higher scores are indicative of better restorative sleep.
Change in Sleep Depth Question (SDQ) Score | baseline, visit 3 (week 1), visit 4 (week 1), visit 5 (week 2), visit 6 (week 2), visit 7 (week 3), visit 8 (week 3), visit 9 (week 4), visit 10 (week 4)
  Participants will be asked to rate the depth of their prior night's sleep using 5-point Likert-type scale. How deep was your sleep? from 1 (light) to 5 (deep) after every sleep laboratory visit.
Change in Pittsburgh Sleep Quality Index (PSQI) Score | baseline, post-intervention (week 5)
  This validated questionnaire evaluates subjective sleep quality. Each of the questionnaire's 19 self-reported items belongs to one of seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Five additional questions rated by the respondent's roommate or bed partner are included for clinical purposes and are not scored. Each component is scored 0 (no difficulty) to 3 (severe difficulty), scores ranging from 0 to 21. Higher scores are indicative of worse sleep quality.
Change in Suicide Risk Survey | baseline, post-intervention (week 5)
  This battery assesses known suicide risk factors. The 13 items ask participants about their sociodemographic characteristics; past experiences with mental health symptoms; thoughts of self-harm, and self-harming actions; psychological traits. Scores range from < 0.39408955691660219 to >= 0.67215170692043313 with higher scores indicative of increased suicidality.
Change in Brief Suicide Cognitions Scale (B-SCS) Score | baseline, post-intervention (week 5), follow-up (week 20)
  This self-report measure assesses the suicide belief system. Using a 5-point likert scale, participants rate 6 items measuring their enduring or identity-based hopelessness rooted in their beliefs about being undesirable, their emotional state as intolerable, and life challenges as insurmountable. Scores range from 6 to 30 where higher scores are indicative of increased suicidality.
Change in Passive and Active Suicidal Ideation Scale (PASIS) Score | baseline, post-intervention (week 5), follow-up (week 20)
  This 17-item validated tool assesses participants' passive and active suicidal ideation in the past seven days using a six-point Likert scale, from 0 (Not in the past 7 days) to 5 (several times every day). Higher score reflects greater suicidal ideation.
Change in NIH Toolbox Loneliness Score | baseline, visit 3 (week 1), visit 4 (week 1), visit 5 (week 2), visit 6 (week 2), visit 7 (week 3), visit 8 (week 3), visit 9 (week 4), visit 10 (week 4), post-intervention (week 5), follow-up (week 20)
  The NIH Toolbox Loneliness consists of 5 self-report items assessing participants' feelings of loneliness and social isolation on a 5-point Likert scale ranging from 1-5 where higher scores indicate increased loneliness.
Change in Five Facet Mindfulness Questionnaire (FFMQ) Score | baseline, visit 3 (week 1), visit 4 (week 1), visit 5 (week 2), visit 6 (week 2), visit 7 (week 3), visit 8 (week 3), visit 9 (week 4), visit 10 (week 4), post-intervention (week 5), follow-up (week 20)
  The FFMQ is a widely used self-report inventory that assesses mindfulness across five facets: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. Participants rate their agreement level with 39 items using a 5-point Likert scale. Scores range from 39 to 195 with higher scores indicative of increased mindfulness.
Change in Drexel Defusion Scale (DDS) Score | baseline, visit 3 (week 1), visit 4 (week 1), visit 5 (week 2), visit 6 (week 2), visit 7 (week 3), visit 8 (week 3), visit 9 (week 4), visit 10 (week 4), post-intervention (week 5), follow-up (week 20)
  This self-report measure evaluates the ability to create a mental separation or distance from one's internal experiences by asking participants to rate 10 items assessing defusion across a spectrum of internal thoughts and emotions on a 6-point scale, ranging from 0-5. Total scores range from 0 to 50 with higher scores indicative of increased defusion.
Change in PROMIS Meaning and Purpose Score | baseline, visit 3 (week 1), visit 4 (week 1), visit 5 (week 2), visit 6 (week 2), visit 7 (week 3), visit 8 (week 3), visit 9 (week 4), visit 10 (week 4), post-intervention (week 5), follow-up (week 20)
  This is a 37-item inventory asks participants to rate their sense of life with purpose and perceived reasons for living using a 5-point Likert scale. The current study will administer the computer adaptive test (CAT) version of the instrument, in which subsequent item choice of the system will be based on participants' previous responses. Scores range from 37 to 185 with higher scores indicative of higher feelings of meaning and purpose.
Change in Digital Working Alliance Inventory (D-WAI) Score | post-intervention (week 5), follow-up (week 20)
  The inventory consists of 6 items which measures the quality of the therapeutic alliance between a user and a digital mental health intervention, which is the HMP in this study. Participants rate their experience using the HMP on a 7-point scale, ranging from 1 (strongly disagree) to 7 (strongly agree). Scores range from 6 to 42 where higher scores indicate better user experience with the app.
Change in Perseverative Thinking Questionnaire (PTQ) Score | baseline, post-intervention (week 5), follow-up (week 20)
  The PTQ is a self-report instrument assessing repetitive and uncontrolled thinking by asking participants to rate 15 items about the frequency, duration, and perceived uncontrollability of repetitive thoughts on a scale of 0-4. Scores range from 0 to 60. The higher the score, the higher the level of perseverative thinking or repetitive thoughts experienced by the individual.
Change in Experiences Questionnaire's Decentering subscale (EQ-D) Score | baseline, post-intervention (week 5), follow-up (week 20)
  This subscale is an 11-item scale of decentering originally developed to assess mechanisms of Mindfulness Based Cognitive Therapy (e.g., "I can separate myself from my thoughts and feelings."). The EQ-D is originally scored on a 5-point Likert scale (1 = never to 5 = all the time) where higher scores indicate increased decentering.
Change in Experience Sampling / Ecological Momentary Assessment | 6 times per day for 7 days
  The experience sampling method assesses present moment experience using a short series of questions administered on a smart phone 6 times a day for 7 days. Questions measure current emotional and cognitive state. Score range from 1-5 where higher scores indicate increased emotional state
Change in Death Implicit Association Test Score | baseline, post intervention (5 weeks)
  This task involves participants viewing words on a screen. Words are either related to self (e.g., "I"), others (e.g., "They"), life (e.g., "survive") or death (e.g., "die"). Like other Implicit Association Tests, participants are asked to indicate which category each word belongs to. Across the trials, self and other are paired with either life or death. The measure can be scored as an implicit marker of how easily participants associated death with themselves. Scores are greater than 2 or less than 2, with more positive values indicating a stronger association between self and death.
Change in Reversal Learning Task Score | baseline, post intervention (5 weeks)
  This task involves participants viewing and choosing between two abstract visual stimuli (i.e., geometric shapes). After each choice they receive feedback that is either positive (+10) or negative (-10) feedback devoid of monetary value. Stimulus-outcome pairings are reversed over the course of the experiment.
Change in Multi-Source Interference Task Score | baseline, post intervention (5 weeks)
  This task involves viewing a series of numbers and letters. Participants are asked to indicate using a button press which number was different from the other numbers. Scores are reported as percentage correct.
Change in Emotional Stroop Score: Reaction Time | baseline, post intervention (5 weeks)
  This task involves viewing a series of faces and words. Participants are asked to identify the emotional expression of the faces. Percent change in reaction time is reported.
Change in Emotional Stroop Score: Percent Correct | baseline, post intervention (5 weeks)
  This task involves viewing a series of faces and words. Participants are asked to identify the emotional expression of the faces. Percent correct is reported.
Change in Meteor Mission Score: Mean Reaction Time | baseline, post-intervention (week 5), follow-up (week 20)
  This is a mobile measure of attention, based on the Sustained Attention to Response Task (SART), a validated, standardized laboratory task. This task lasts five minutes and measures attention regulation and sustained attention, as assessed based on reaction time, reaction time variability, and accuracy.
Change in Meteor Mission Score: Coefficient of Variation | baseline, post-intervention (week 5), follow-up (week 20)
  This is a mobile measure of attention, based on the Sustained Attention to Response Task (SART), a validated, standardized laboratory task. This task lasts five minutes and measures attention regulation and sustained attention, as assessed based on reaction time, reaction time variability, and accuracy.
Change in Meteor Mission Score: Percent Correct | baseline, post-intervention (week 5), follow-up (week 20)
  This is a mobile measure of attention, based on the Sustained Attention to Response Task (SART), a validated, standardized laboratory task. This task lasts five minutes and measures attention regulation and sustained attention, as assessed based on reaction time, reaction time variability, and accuracy.
Change in Emotional Persistence Task Score | baseline, post intervention (5 weeks)
  This task involves viewing pictures categorized as neutral, positive, or negative. Participants may be asked to press a button indicating the valence category of the picture. Positive and negative affect ratings will be made on a continuous sliding scale ranging from 0 to 6.
Change in Change Your Mind Task Score: Mean Change | baseline, post intervention (5 weeks)
  This task involves viewing a series of letters and numbers. Participants are asked to determine whether a target letter was a certain letter (e.g., "T"). Participants receive feedback on their choices. The feedback is not always accurate and participants are informed of this. Change range is from 0 to 1.
Change in Change Your Mind Task Score: Accuracy | baseline, post intervention (5 weeks)
  This task involves viewing a series of letters and numbers. Participants are asked to determine whether a target letter was a certain letter (e.g., "T"). Participants receive feedback on their choices. The feedback is not always accurate and participants are informed of this. Accuracy is from 0 to 1.
Change in Change Your Mind Task Score: Response Time | baseline, post intervention (5 weeks)
  This task involves viewing a series of letters and numbers. Participants are asked to determine whether a target letter was a certain letter (e.g., "T"). Participants receive feedback on their choices. The feedback is not always accurate and participants are informed of this. Response time is reported.
Psychomotor Vigilance Task (Phase 2 only) | baseline, visit 3 (week 1), visit 4 (week 1), visit 5 (week 2), visit 6 (week 2), visit 7 (week 3), visit 8 (week 3), visit 9 (week 4), visit 10 (week 4)
  Psychomotor vigilance performance will be measured with the visual psychomotor vigilance task (PVT) a portable, easily usable reaction-time test with a that can yield rapid and reliable assessments of psychomotor vigilance impairment. Participants will take a 3 minute version of the PVT on a tablet or laptop every morning after an in-laboratory sleep visit to assess alertness. Reaction time is reported.

SECONDARY OUTCOMES:
Change in Spectral Power Density During Stimulation-Free Sleep | baseline and up to 8 nights (4 nights for the low frequency group) over the 4 week intervention period following the baseline assessment
  Change in individual participant spectral power density during stimulation free sleep will be measured and reported separately for NREM sleep (in the 1-4 Hz frequency range) and REM sleep (in the approximately 50hz frequency range) at circadian time-matched periods of baseline sleep and time-matched, stimulation free periods on each of the intervention nights.
Resting-state fMRI Connectivity Z-Scores | baseline, post intervention (5 weeks)
  Resting-state fMRI connectivity will be assessed based on the Fisher-Z transformed (FZT) correlation of each seed region with all other voxels in the brain. In order to test for intervention effects, difference maps will be computed and a voxelwise analysis of the difference maps across the whole brain will be used to identify regions that might differ in connectivity between groups over time. A z-score is the number of standard deviations away from the mean.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Davidson, PhD, Principal Investigator — University of Wisconsin, Madison; Giulio Tononi, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Center for Healthy Minds, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be kept for an indefinite period. Banked data will be kept in a secure location for use by researchers. The data may be shared with other researchers at the University of Wisconsin-Madison and outside the University. Outside researchers may be at other universities, private companies, or other kinds of organizations. The banked data will be labeled with a code instead of a participant's name. When the data is shared with other investigators for research projects, they will not be able to use the code to figure out which data belongs to a particular subject. The research team will maintain a link between the data and subject identifiable information kept by the study team. This link will not be shared with anyone outside of the study team. Participants will be able to request to have their data removed from the bank by contacting the research team at any time.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Data sharing will be available by request and will be granted on an individual basis. In addition, fully de-identified data will be shared for open access purposes.

REFERENCES:
- See also: Center for Healthy Minds — https://centerhealthyminds.org/